CLINICAL TRIAL: NCT05689632
Title: Effects of Vitamin D3 and Vitamin K2MK7 Supplementation on Vascular Function in Overweight or Obese Adults.
Brief Title: Vitamins D and K Effects on Vascular Function in Obese Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Mario Fritsch Neves, FULL PROFESSOR, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CVH-D3K2
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Vitamin D3 Deficiency
Keywords: Obesity; Vitamin D3 Deficiency; Vitamin K; Sympathetic tonus; Endothelial dysfunction; Arterial stiffness
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, double-blind study
Who Masked: Outcomes Assessor
Masking Description: The participants and the investigator do not know which supplements are taken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo - Medium-chain triglyceride
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 (Active Comparator): Vitamin D3 - 7000 IU daily
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 + K2-MK7 (Experimental): Vitamin D3 - 7000 IU + Vitamin K2-MK7 180mcg combined, daily
  Interventions: Dietary Supplement: Vitamin D3 + K2-MK7

INTERVENTIONS:
Dietary Supplement: Vitamin D3 + K2-MK7 — Combined supplementation
  Arms: Vitamin D3 + K2-MK7
Dietary Supplement: Placebo — MCT
  Arms: Placebo
Dietary Supplement: Vitamin D3 — Vitamin D3 - 7000 IU
  Arms: Vitamin D3

SUMMARY:
A prospective, randomized, placebo-controlled, double-blind study that aims to evaluate the effects of combined vitamin D3 and K2-MK7 supplementation on vascular function, sympathetic tone, metabolic biomarkers and inflammatory factors in a population of overweight or obese adults and deficient or insufficient serum levels of vitamin D.

DETAILED DESCRIPTION:
Overweight and obesity are public health issues of epidemic proportions nowadays. They constitute risk factors for several chronic diseases with vascular, metabolic, and inflammatory changes. Adequate serum levels of vitamin D are correlated with good cardiovascular and metabolic health, since its deficiency and insufficiency (highly prevalent in obesity) have an inverse correlation. Likewise, vitamin K, especially K2, is related to the reduction of arterial stiffness, suppression of the inflammation in the vascular wall, favorable action on the lipid profile, whereas insufficiency is related to increased cardiovascular risk. The combined use of vitamin D and K aiming to reduce cardiovascular risk has been studied, however, the results of randomized clinical trials are still controversial. This prospective, randomized, placebo-controlled, double-blind trial aims to evaluate the effect of supplementation of vitamins D3 and K2-MK7 on vascular function, sympathetic tone, metabolic biomarkers and inflammatory factors in a population of overweight or obese adults and serum levels of deficient or insufficient vitamin D. Individuals of both sexes, aged between 40 and 70 years, body mass index (BMI) ≥ 25 and < 40 kg/m² and vitamin 25OHD3 <30 ng/ml will be randomized into 3 groups (A/B/C) to receive supplementation (Placebo/VitD3 7000 IU/VitD3 7000IU+K2-MK7-180mcg) daily for 16 weeks. Individuals will be rated at 4 visits namely:

* V0 screening according to inclusion and exclusion criteria; clinical, anthropometry and electrical bioimpedance, laboratory and vascular evaluation before supplementation;
* V1 supplementation begins;
* V2 after 8 weeks;
* V3 at the end of the intervention. The laboratory evaluation consists of blood count, biochemistry, electrolytes, glucose, lipid, liver and thyroid profiles, vitamin D3 and parathyroid hormone, in addition to the urinary excretion of calcium and creatinine. Sympathetic tone is assessed by a frequency meter (Polar® Verity Sense), arterial stiffness by measuring the pulse wave velocity by oscillometry (Mobil-O-Graph®) and endothelium function by measuring post-occlusion microvascular reactivity using laser speckle contrast image-LSCI.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D deficiency;
* Vitamin D insufficiency;
* Obesity;
* Overweight;

Exclusion Criteria:

* Diabetes mellitus;
* Arterial coronary disease;
* Beta blocker use;
* cancer;
* ESRD;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Microvascular reactivity | 150 minutes
  A laser speckle contrast imaging system with a laser wavelength of 785 nm system will measure non-invasively real time cutaneous microvascular flow changes in the forearm. For the post occlusive reactive hyperemia test, arterial occlusion will be performed with suprasystolic pressure (50 mmHg above the systolic arterial pressure) using a sphygmomanometer applied to the arm of the subject over three minutes. Peak skin flow will be measured after pressure release.

SECONDARY OUTCOMES:
Central blood pressure | 150 minutes
  Central systolic blood pressure, diastolic blood pressure, mean arterial pressure and pulse pressure before and after intervention and their potential effects on changes in subendocardial viability ratio and ejection duration after intervention with beetroot juice and water.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana C Faria, MD, Principal Investigator — State University of Rio de Janeiro; Mario F Neves, MD, PhD, Study Director — State University of Rio de Janeiro
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD with other researchers